CLINICAL TRIAL: NCT03970395
Title: Effectiveness of Osteopathic Manipulative Therapy in Nonsynostotic Plagiocephaly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PRIOLO CLAUDIO (Other)
Collaborators: Scuola Superiore di Osteopatia Italiana (Other)
Responsible Party: Sponsor-Investigator, PRIOLO CLAUDIO, Paediatrician, A.O.U. Città della Salute e della Scienza
Organization: A.O.U. Città della Salute e della Scienza (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0074260
Record Dates: First submitted 2019-05-05; First posted 2019-05-31 (Actual); Results first posted 2020-09-24 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Nonsynostotic Plagiocephaly
Keywords: Positional Plagiocephaly, Deformational Plagiocephaly,
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: A two arms randomized controlled trial. The experimental group will receive Osteopathic manipulative Therapy and the active comparator the Light Touch Therapy
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Infants were randomly assigned to two groups, OMT and LTT by using a random number generator, prepared in advance by an independent biostatistician. Sequentially numbered, opaque, and sealed envelopes were used.
  Clinician-Investigators, neonatology staff, the physical therapist, and the osteopath in charge of assessment were unaware of the random list.
  Infants' parents, after having signed the informed consent form, chose the numbered envelope and were unaware of the random list for the whole period of study.
  The two osteopaths in charge of Osteopathic manipulative therapy and Light Touch Therapy were unblinded to group assignment.
  Clinical outcomes were assessed by a biostatistician who was not involved in the patients' clinical allocation and management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic manipulative therapy (Experimental): Repositioning Therapy plus Osteopathic Manipulative Therapy (OMTh).
  Osteopathic Manipulative Therapy. Participant OMT group receive 6 OMTh in 3 months, as follows: first at baseline, the second after 1 week, the third after 3 weeks, and then once every 3 weeks for three more visits.
  Interventions: Other: Osteopathic manipulative therapy (OMTh); Other: Repositioning therapy
- Light Touch Therapy (Sham Comparator): Repositioning Therapy plus Light Touch Therapy (LTT)
  Participants to the LTT group receive the LTT protocol at the same date of the OMTh group.
  Interventions: Other: Light Touch Therapy (LTT); Other: Repositioning therapy

INTERVENTIONS:
Other: Osteopathic manipulative therapy (OMTh) — The Osteopathic Manipulative Therapy includes evaluation and treatment. The evaluation considers the pelvic girdle and lower limb, thorax abdominal area, pectoral girdle and upper limbs, cervical and upper thoracic area, cranial vault, cranial base and viscero cranium. The treatment is based on balanced ligamentous tension technique, myofascial release, visceral manipulation, and balanced membranous tension technique. The OMTh lasts for 45 minutes of which 15 minutes of evaluation and 30 minutes of treatment.
  Arms: Osteopathic manipulative therapy
Other: Light Touch Therapy (LTT) — The LTT is consistent with the OMT during the phase of evaluation. The treatment retains the same areas used for osteopathic approach but avoids prolonged touch in any area of the body, moving the hands every few seconds, and by flattening and softening the surface of the hands to minimize focal areas of force.
  Arms: Light Touch Therapy
Other: Repositioning therapy — It consists of strategies that guide the parents to position the baby "back to sleep", by alternating head position, the use of tummy time while supervised, and the infants must spend minimal time in car seats or other devices that promote supine positions. In active counter-positioning the parents are suggested to place some toys on the side of the head where neck rotation is limited while, when using the changing table, to alternate the end of the table at which the infant's head is placed.

SUMMARY:
The aim of this trial is to evaluate the effectiveness of osteopathic manipulative therapy in reducing the asymmetries of skull in infants with nonsynostotic plagiocephaly.

DETAILED DESCRIPTION:
Nonsynostotic plagiocephaly (NSP) is defined as the deformation of the head resulting from external forces that mould the skull during the first months of life.

Four months seems to be a critical age for the development of NSP, but many positional head shape deformities may improve with time.

Early assessment and diagnosis is important not only for the shape of the skull, but also for possible clinical significant differences in gross motor development.

In paediatric conditions the effect of osteopathic manipulative treatment is documented in systematic reviews; in NSP the only study, which is a pilot, reveals an average reduction of 50% asymmetry on 12 infants who have undergone a course of four osteopathic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Infants with NSP, ODDI score of 104% or more.
* To be at term corrected age if born prematurely.

Exclusion Criteria:

* Synostotic Plagiocephaly
* Infant who underwent an osteopathic manipulative treatment before the enrolment
* Dysmorphisms
* Syndromes
* Congenital Muscular Torcicolis
* Cerebral Palsy

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G Priolo, Medical, Study Director — Azienda Ospedaliera Città della Salute e della scienza di Torino _ Italy; Daniele Farina, Medical, Principal Investigator — Azienda Ospedaliera Città della Salute e della scienza di Torino _ Italy
Locations (1):
- Division of Neonatology and NICU, Sant'Anna Hospital, Azienda Ospedaliera Universitaria Città della Salute e della Scienza., Torino, Italy

REFERENCES:
- [Background] Rogers GF. Deformational plagiocephaly, brachycephaly, and scaphocephaly. Part I: terminology, diagnosis, and etiopathogenesis. J Craniofac Surg. 2011 Jan;22(1):9-16. doi: 10.1097/SCS.0b013e3181f6c313. PMID 21187783
- [Background] Rogers GF. Deformational plagiocephaly, brachycephaly, and scaphocephaly. Part II: prevention and treatment. J Craniofac Surg. 2011 Jan;22(1):17-23. doi: 10.1097/SCS.0b013e3181f6c342. PMID 21187782
- [Background] Lennartsson F. Developing guidelines for child health care nurses to prevent nonsynostotic plagiocephaly: searching for the evidence. J Pediatr Nurs. 2011 Aug;26(4):348-58. doi: 10.1016/j.pedn.2010.07.003. Epub 2010 Sep 25. PMID 21726785
- [Background] Lessard S, Gagnon I, Trottier N. Exploring the impact of osteopathic treatment on cranial asymmetries associated with nonsynostotic plagiocephaly in infants. Complement Ther Clin Pract. 2011 Nov;17(4):193-8. doi: 10.1016/j.ctcp.2011.02.001. Epub 2011 Mar 5. PMID 21982132
- [Background] van Vlimmeren LA, Takken T, van Adrichem LN, van der Graaf Y, Helders PJ, Engelbert RH. Plagiocephalometry: a non-invasive method to quantify asymmetry of the skull; a reliability study. Eur J Pediatr. 2006 Mar;165(3):149-57. doi: 10.1007/s00431-005-0011-1. Epub 2005 Oct 7. PMID 16211401
- [Derived] Bagagiolo D, Priolo CG, Favre EM, Pangallo A, Didio A, Sbarbaro M, Borro T, Dacco S, Manzoni P, Farina D. A Randomized Controlled Trial of Osteopathic Manipulative Therapy to Reduce Cranial Asymmetries in Young Infants with Nonsynostotic Plagiocephaly. Am J Perinatol. 2022 Dec;39(S 01):S52-S62. doi: 10.1055/s-0042-1758723. Epub 2022 Nov 30. PMID 36451623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 129 infants screened at Sant'Anna Hospital, 96 were enrolled between September 2016 and June 2019.
Groups:
- Osteopathic Manipulative Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Osteopathic Manipulative Therapy (OMTh).
  They received 6 OMTh in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention were performed by two osteopath with specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
- Light Touch Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Light Touch Therapy (LTT).
  They received 6 LTT in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention were performed by two osteopath with specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
Period: Overall Study
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Started | 48 | 48
Completed | 41 | 36
Not Completed | 7 | 12
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Osteopathic Manipulative Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, Oblique Diameter Difference Index (ODDI )score >= 104% were randomized to Repositioning Therapy plus Osteopathic Manipulative Therapy (OMTh).
  They received 6 OMTh in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
- Light Touch Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, Oblique Diameter Difference Index (ODDI) score >= 104% were randomized to Repositioning Therapy plus Light Touch Therapy (LTT).
  They received 6 LTT in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
- Total: Total of all reporting groups
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: months] | 3.1 (1.4) | 3.2 (1.6) | 3.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 27 | 26 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 48 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 48 | 48 | 96
Gestational Age [Mean (Standard Deviation); unit: weeks] | 36.7 (3.9) | 34.3 (4.6) | 35.5 (4.2)
Presentation at birth [Count of Participants; unit: Participants]
  Cefalic | 39 | 37 | 76
  Breech | 2 | 6 | 8
  Trasvers | 7 | 5 | 12
Birth weight [Mean (Standard Deviation); unit: grams] | 2657 (945) | 2290 (995) | 2473 (970)
Mother's first pregnancy [Count of Participants; unit: Participants] | 24 | 26 | 50
Multiple birth [Count of Participants; unit: Participants] | 6 | 10 | 16
Delivery [Count of Participants; unit: Participants]
  Vaginal | 14 | 11 | 25
  Assisted | 9 | 6 | 15
  Vacuum - Forceps | 4 | 4 | 8
  Cesarean | 21 | 27 | 48
Feeding [Count of Participants; unit: Participants]
  Maternal | 14 | 12 | 26
  Bottle | 22 | 26 | 48
  Mix | 12 | 10 | 22
Sleeping [Count of Participants; unit: Participants]
  Supine | 46 | 48 | 94
  Variable | 2 | 0 | 2
Daytime [Count of Participants; unit: Participants]
  Supine | 35 | 34 | 69
  Variable | 13 | 14 | 27
Mother's age [Mean (Standard Deviation); unit: years] | 33.8 (5.4) | 35.1 (6.5) | 34.45 (5.95)
Father's age [Mean (Standard Deviation); unit: years] | 36.9 (6.8) | 37.1 (6.8) | 37 (6.8)
Age end of study [Mean (Standard Deviation); unit: months] | 6.1 (1.4) | 6.2 (1.6) | 6.15 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change From Baseline in ODDI Score (Oblique Diameter Difference Index) to Below 104% at 3 Months
Description: The ODDI score being the most clinically relevant measure to define nonsynostotic plagiocephaly.
  The category of nonsynostotic plagiocephaly is defined by reference to the following score:
  ODDI score >=104 Nonsynostotic Plagiocephaly ODDI score <104 Absence of Nonsynostotic Plagiocephaly Higher score means a worse outcome.
Time Frame: Baseline and 3 months
Population: Intent to Treat Population (all infants assigned to OMTh or LTT). Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Groups:
- Osteopathic Manipulative Therapy Plus Repositioning Therapy: Participants received Osteopathic Manipulative Therapy (OMTh) plus Repositioning Therapy.
  OMTh: 6 treatments in 3 months, first at baseline, second at 1 week, third at 3 weeks, and then 3 more at 3 weeks.
- Light Touch Therapy Plus Repositioning Therapy: Participants received Light Touch Therapy (LTT) plus Repositioning Therapy. LTT: 6 treatments in 3 months, first at baseline, second at 1 week, third at 3 weeks, and then 3 more at 3 weeks.
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 48 | 48
Participants
  ODDI score <104% | 23 | 3
  ODDI score >=104% | 25 | 45
Statistical Analysis 1: Comparison: Osteopathic Manipulative Therapy Plus Repositioning Therapy vs Light Touch Therapy Plus Repositioning Therapy; Test type: Superiority; p = 0.01, Risk Ratio (RR) — The threshold for statistical significance was p<0.5; Risk Ratio (RR) = 7.66, 95% CI 2-sided [2.46 to 23.84] — Risk Difference 0.41 (IC 95; 0.25-0.53)

2. Primary Outcome: Number of Participants With Change From Baseline in ODDI Score (Oblique Diameter Difference Index) to Below 104% at 1 Year of Age.
Description: as for outcome 1
Time Frame: Follow-up at 1 year of age
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Osteopathic Manipulative Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Osteopathic Manipulative Therapy (OMTh).
  They received 6 OMTh in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention were performed by two osteopaths with specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
- Light Touch Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Light Touch Therapy (LTT).
  They received 6 LTT in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention were performed by two osteopaths with specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 48 | 48
Participants
  ODDI score <104% | 28 | 5
  ODDI score >=104% | 20 | 43
Statistical Analysis 1: Comparison: Osteopathic Manipulative Therapy Plus Repositioning Therapy vs Light Touch Therapy Plus Repositioning Therapy; Test type: Superiority; p = 0.01, Relative Risk (RR); Risk Ratio (RR) = 5.6, 95% CI 2-sided [2.36 to 13.27] — Risk Difference 0.47 (IC 95; 0.31-0.64)

3. Primary Outcome: Number of Participants With Change From Baseline in ODDI Score (Oblique Diameter Difference Index) to Below 104% at 3 Months
Description: as for outcome 1
Time Frame: At 3 months
Population: Per Protocol population, defined as participants completing the three months intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 45 | 44
Participants
  ODDI score <104% | 23 | 3
  ODDI score >=104% | 22 | 41
Statistical Analysis 1: Comparison: Osteopathic Manipulative Therapy Plus Repositioning Therapy vs Light Touch Therapy Plus Repositioning Therapy; Test type: Superiority; p = 0.01, Risk Ratio (RR); Risk Ratio (RR) = 7.49, 95% CI 2-sided [2.42 to 23.18] — Risk Difference 0.44 (IC 95%; 0.27-0.60)

4. Primary Outcome: Number of Participants With Change From Baseline in ODDI Score (Oblique Diameter Difference Index) to Below 104% at 1 Year of Age.
Description: The ODDI score being the most clinically relevant measure to define nonsynostotic plagiocephaly.
  The category of Nonsynostotic plagiocephaly is defined by reference to the following score:
  ODDI score >=104<108 MILD Nonsynostotic Plagiocephaly ODDI score >=108<112 MODERATE Nonsynostotic Plagiocephaly ODDI score >= 112 SEVERE Nonsynostotic Plagiocephaly Higher score means a worse outcome.
Time Frame: Follow-up at one year of age
Population: Per Protocol population, defined as participants completing the one year of age follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 41 | 36
Participants
  ODDI score <104% | 28 | 5
  ODDI score >=104% | 13 | 31
Statistical Analysis 1: Comparison: Osteopathic Manipulative Therapy Plus Repositioning Therapy vs Light Touch Therapy Plus Repositioning Therapy; Test type: Superiority; p = 0.01, Risk Ratio (RR); Risk Ratio (RR) = 4.91, 95% CI 2-sided [2.12 to 11.38] — Risk Difference 0.54 (IC 95; 0.36-0.72)

5. Secondary Outcome: Cranial Proportion Index (CPI)
Description: Change of the width and length diameter measured with Plagiocephalometry.
Time Frame: The change of CPI will be measured at baseline, at 3 months from baseline and follow-up at 1 year of age.
Population: Data were not collected for lack of clinical relevance
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Event
Description: Symptoms such as irritability accured after the Osteopathic Manipulative Therapy or Light Touch Therapy
Time Frame: From first treatment (1 week post-baseline) up to end of treatment course (3 months).
Population: Any Adverse Events
Measure: Count of Participants; unit: Participants
Groups:
- Osteopathic Manipulative Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Osteopathic Manipulative Therapy (OMTh).
  They received 6 OMTh in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention were performed by two osteopaths with a specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
- Light Touch Therapy Plus Repositioning Therapy: Participants with Nonsynostic Plagiocephaly, ODDI score >= 104% were randomized to Repositioning Therapy plus Light Touch Therapy (LTT).
  They received 6 LTT in 3 months, as follows: first at baseline, second after 1 week, third after 3 weeks, and then three more visits every 3 weeks.
  The intervention was performed by two osteopaths with a specific background in paediatric field.
  Repositioning therapy: It consists of strategies that guide the parents to position the baby "back to sleep".
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
Number analyzed (Participants) | 48 | 48
Participants
  Serious Adverse events | 0 | 0
  Other adverse events such as irritability | 0 | 0

ADVERSE EVENTS:
Time Frame: From first treatment (1 week post-baseline) up to end of treatment course (3 months).
Description: Symptoms such as irritability occured after the Osteopathic Manipulative Therapy or Light Touch Therapy
Arm/Group | Osteopathic Manipulative Therapy Plus Repositioning Therapy | Light Touch Therapy Plus Repositioning Therapy
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT03970395/Prot_SAP_000.pdf